CLINICAL TRIAL: NCT04080349
Title: Comparison of Vaginal Misoprostol and Dinoprostone Prior to Copper Intrauterine Device Insertion in Women Delivered Only by Cesarean Delivery:a Randomized Controlled Trial
Brief Title: Comparison of Vaginal Misoprostol and Dinoprostone Prior to Copper Intrauterine Device Insertion in Women Delivered Only by Cesarean Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dinoprostone misoprostol IUDs
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: IUD Pain
MeSH Terms: interventions — Dinoprostone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dinoprostone (Experimental): 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 3 hours before IUD insertion.
  Interventions: Drug: Dinoprostone 3 mg
- misoprostol (Active Comparator): 1 vaginal tablet of misoprostol (200 mcg) (Misotac®; Sigma Pharma, SAE, Egypt) inserted by the study nurse 3 hours before IUD insertion.
  Interventions: Drug: Misoprostol 200Mcg Tab
- placebo (Placebo Comparator): one tablet of placebo inserted by the study nurse 3 hours before IUD insertion.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dinoprostone 3 mg — 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 3 hours before IUD insertion.
  Arms: dinoprostone
Drug: Misoprostol 200Mcg Tab — 1 vaginal tablet of misoprostol (200 mcg) (Misotac®; Sigma Pharma, SAE, Egypt) inserted by the study nurse 3 hours before IUD insertion.
  Arms: misoprostol
Drug: placebo — one tablet of placebo inserted by the study nurse 3 hours before IUD insertion
  Arms: placebo

SUMMARY:
To compare the effect of vaginal dinoprostone versus vaginal misoprostol administered before the copper intrauterine device(IUD) insertion in reducing IUD insertion pain and the difficulty in inserting the IUD in women delivered only by cesarean section.

DETAILED DESCRIPTION:
Long-acting reversible contraception methods are highly effective methods for reduction of the unplanned pregnancy rate worldwide. The intrauterine device is a single procedure that provides reliable, effective and long term contraception for many women. However, the insertion procedure can be associated with a troublesome degree of pain that prevent some women from choosing its use. Different interventions have been described to decrease pain perception during intrauterine device insertion with no agreement on an effective one.

ELIGIBILITY:
Inclusion Criteria:

* women delivered only by elective cesarean section and not received analgesics in the last 24 hours

Exclusion Criteria:

* contraindications to dinoprostone or misoprostol or IUD insertion and allergy to study drugs.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-09-10 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-05 (Estimated)

PRIMARY OUTCOMES:
The difference in pain scores during intrauterine device insertion | 10 minutes
  The difference in pain scores during intrauterine device insertion using visual analog scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University